CLINICAL TRIAL: NCT03321669
Title: Impact of Diet on Capsule Endoscopy Transit Time - a Pilot Study
Brief Title: Impact of Diet on Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Britanico (Other)
Responsible Party: Principal Investigator, Juan Sebastian Lasa, Principal Investigator, Hospital Britanico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HB764
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Small Bowel Disease
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Increased Fat Diet (Active Comparator)
  Interventions: Procedure: Capsule endoscopy
- Low Fat Diet (Sham Comparator)
  Interventions: Procedure: Capsule endoscopy

INTERVENTIONS:
Procedure: Capsule endoscopy — Ingestion of capsule endoscopy for the diagnosis of small bowel lesions

SUMMARY:
Capsule endoscopy studies are used for the diagnosis of small bowel mucosal lesions. Since capsule endoscopy depends on the small intestinal peristaltism, the food intake - especially the amount of fat ingested - after the ingestion of the capsule may have an impact on the capsule endoscopy transit time and thus its diagnostic yield. As a consequence, an open-label randomized pilot study was designed to determine wether increased dietary intake of fat after the ingestion of the capsule endoscopy may influence small intestinal transit time and thus the diagnosis of small bowel lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing capsule endoscopy study

Exclusion Criteria:

* Not being able to follow a diet with increased amount of fat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Small bowel transit time | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Britanico, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided